CLINICAL TRIAL: NCT02638038
Title: A 6-month, Double-blind, Randomized, Parallel-group, Multicenter Study Comparing Safety and Efficacy of Monotherapy With INT131 1 mg or 3 mg or Placebo Administered Orally Once Daily in Treatment Naïve Patients (Who Never Received Disease Modifying Treatment) With Relapsing-Remitting Multiple Sclerosis
Brief Title: This is a Randomized Study Comparing Two Doses of INT131 ( 3 mg and 1 mg) Administered Orally (PO) Daily (QD) Versus Placebo 1 Tablet PO QD in Subjects With Treatment-naïve RRMS for ≤ 3 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InteKrin Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INT131-RU01-2
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — INT 131

STUDY DESIGN:
Intervention Model Description: A randomized double blind parallel group study with 3mg, 1mg or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oral INT 131 3 mg (Experimental): Oral INT-131 Double blind study
  Interventions: Drug: INT131
- Oral INT-131 1 mg (Experimental): Oral INT-131 Double blind
  Interventions: Drug: INT131
- Placebo (Placebo Comparator): Oral placebo Double blind
  Interventions: Drug: INT131

INTERVENTIONS:
Drug: INT131 — INT- 131

SUMMARY:
This is a randomized, double-blind, parallel group study comparing two doses of INT131( 3 mg and 1 mg) administered orally (PO) daily (QD) versus placebo 1 tablet PO QD in subjects with treatment-naïve RRMS for ≤ 3 years.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group study comparing two doses of INT131( 3 mg and 1 mg) administered orally (PO) daily (QD) versus placebo 1 tablet PO QD in subjects with treatment-naïve RRMS for ≤ 3 years..

Part 2 of the study is open-label, Subjects completing 6 months of evaluations and study drug in Part 1 without serious study drug-related treatment emergent adverse events (TEAE) will be switched to INT131 1 mg PO QD and followed for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before any study procedures
2. Male and female subjects aged 18-50
3. Subjects with a diagnosis of RRMS of three (3) years or less based on date of diagnosis
4. At least one gadolinium-positive lesion within twelve months of enrollment in the study documented in subject's clinical chart

Exclusion Criteria:

1. Subjects with a history or presence of chronic disease of the immune system other than RRMS
2. Subjects with a diagnosis of primary or secondary progressive multiple sclerosis
3. Ten (10) or more active gadolinium CE MRI-detected lesions on baseline MRI obtained on visit 2

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2016-12-12 (Actual)

PRIMARY OUTCOMES:
The number of new gadolinium CE T1 weighted lesions | asline to 6 months
  The mean number of new gadolinium CE T1-weighted lesions, on monthly MRI in subjects receiving INT131 compared to Placebo from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K. Finck, M.D, Study Chair — Coherus BioSciences (parent company for Zao InteKrin)